CLINICAL TRIAL: NCT04448223
Title: Multi Center, Randomized, Open-label, Active Controlled, Phase 2 Trial, Proof Of Concept Study to Evaluate the Efficacy and Safety of CKD-351 in Primary Open Angle Glaucoma or Ocular Hypertension Patients
Brief Title: A Clinical Study to Evaluate the Efficacy and Safety of CKD-351
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: A71_04GLC1915
Record Dates: First submitted 2020-05-11; First posted 2020-06-25 (Actual); Last update posted 2020-06-25 (Actual); Status verified 2020-06

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary Open-angle Glaucoma; Ocular Hypertension; CKD-351
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CKD-351 (Experimental): CKD-351
  Interventions: Drug: CKD-351
- Latanoprost+Dorzolamide (Active Comparator): Latanoprost(50ul/ml) Dorzolmamide(20mg/ml)
  Interventions: Drug: Latanoprost+Dorzolmamide

INTERVENTIONS:
Drug: CKD-351 — Latanoprost (25ug/ml), Dorzolamide (20mg/ml), twice a day
  Arms: CKD-351
Drug: Latanoprost+Dorzolmamide — Latanoprost(50ug/ml) , once a day Dorzolmamide(20mg/ml), threetimes a day
  Arms: Latanoprost+Dorzolamide

SUMMARY:
The purpose of this study is to evaluate efficacy and safety of CKD-351

DETAILED DESCRIPTION:
Multi center, Randomized, Open-label, Active controlled, Phase 2 trial, Proof Of Concept Study to evaluate the efficacy and safety of CKD-351 in primary open angle glaucoma or ocular hypertension patients

ELIGIBILITY:
Inclusion Criteria:

1. More than the age of 19 years old
2. Subjects who has primary open-angle glaucoma or ocular hypertension
3. Subjects who sign on an informed consent form willingly

Exclusion Criteria:

1. Subjects with intraocular pressure ≥ 35 mmHg at Visit 1 or Visit 2 (AM 09:00)
2. Subjects with a maximum corrected visual acuity ≤ 0.3 in the selected evaluation eye at Visit 1 or Visit 2
3. Subjects who were diagnosed as below

   * Aphakia
   * Intraocular lens
   * Acute or Chronic Closed-Angle Glaucoma
   * Secondary Glaucoma
4. Subjects with ocular inflammation or infection within the last 3 months
5. Subjects with significant history of ocular trauma during the last 6 months or who underwent surgical opthalmic surgery
6. Subjects who received topical or systemic steroids within the last 1 month.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-06-11 (Actual); Primary Completion 2022-12-05 (Estimated); Study Completion 2022-12-05 (Estimated)

PRIMARY OUTCOMES:
Change in mean intraocular pressure for efficacy measurement | Baseline, 4 weeks
  Change in mean intraocular pressure at 4 weeks compared to baseline

SECONDARY OUTCOMES:
Change in mean intraocular pressure for efficacy measurement | Baseline, 2 weeks
  Change in mean intraocular pressure at 2 weeks compared to baseline
Changes in intraocular pressure for efficacy measurement | Baseline, 2 weeks, 4 weeks
  Intraocular pressure by each measurement time

CONTACTS AND LOCATIONS:
Overall Officials: KiHo Park, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No